CLINICAL TRIAL: NCT04820946
Title: Evolution of Children and Adolescents With Disruptive Mood Dysregulation Disorder Refereed to Hospital for Suicidal Behavior After Three Year: Diagnostic Stability, Psychiatric Comorbidity, Psychosocial Functioning, Identification of Clinical and Actigraphy-measured Prognosis Factors
Brief Title: Evolution of DMDD Children and Adolescent
Acronym: ACTIHUMEURp3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0013
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Disruptive Mood Dysregulation Disorder; Prognosis Factors; Suicidal Behaviors; Actigraphy
Keywords: Disruptive Mood Dysregulation Disorder; prognosis factors; natural course; suicidal behaviors; actigraphy; pediatric depressive disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- various episodic mood disturbances patient group: A group of patients with various episodic mood disturbances was used as a clinical case control group.
- Disruptive Mood Dysregulation Disorder (DMDD) patient group: DMDD patients referred to the hospital for suicidal behaviors between 2013 and 2018 in terms of diagnostic stability, psychiatric comorbidity, and psychosocial factors.

SUMMARY:
Little is known about the natural course and prognosis factors of inpatients and outpatients with Disruptive Mood Dysregulation Disorder (DMDD). The investigators conducted a cross-sectional study to determine the evolution of a sample of DMDD patients referred to the hospital for suicidal behaviors between 2013 and 2018 in terms of diagnostic stability, psychiatric comorbidity, and psychosocial factors. A group of patients with various episodic mood disturbances was used as a clinical case control group.

In addition to change in DMDD symptoms across time, the investigators examined the onset and persistence of psychiatric comorbidity using the KIDDIE-SADS PL and suicidal behaviors using the Colombia Suicidality Severity Rating Scale. The investigators also examined the persistence of depressive symptoms using the Beck Depression Inventory (BDI-II), the persistence of emotional lability (Affective Lability Scale-18), borderline traits (Abbreviated Diagnostic of Inventory Borderline). Socio-demographic, clinical features and actigraphy-measured sleep characteristics determined between 2013 and 2018 were used to predict the evolution of the DMDD patients and the clinical control group.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls between 10 and 25-year-old
* patients who had been referred to the university hospital of Amiens for suicidal behaviors between 2013 and 2018
* patients who participated to the study "Clinical and actigraphy-measured profiles of inpatient youths with suicidal behavior: exploration of the severe mood dysregulation"

Exclusion Criteria:

* No affiliation to a social security service
* Persons deprived of their liberty as stipulated in article L.1121-6 of the Public Health Code

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: DMDD patients referred to the hospital for suicidal behaviors between 2013 and 2018 in terms of diagnostic stability, psychiatric comorbidity, and psychosocial factors.
  A group of patients with various episodic mood disturbances was used as a clinical case control group.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic evolution toward an other psychiatric disorder. | one day
  The evolution toward another psychiatric disorder would be examined using the semi-structured interview KIDDIE-SADS and the Ab-DIB to examine borderline traits.
  The K-SADS is a semi-structured interview to measure current and past symptoms of mood, anxiety, psychotic, and disruptive behavior disorders in children ages 6-18 years old.
  (Ab-DIB) as a screening measure of borderline psychopathology in an adolescent clinical population.
persistence of a full-blown DMDD diagnostic | one day
  The persistence of a full-blown DMDD diagnostic would be defined using the DSM-5 criteria. Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) is the 2013 update to the Diagnostic and Statistical Manual of Mental Disorders, the taxonomic and diagnostic tool published by the American Psychiatric Association.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No